CLINICAL TRIAL: NCT05603169
Title: Effects of High Intensity Resistance and Aerobic Training Among Women With Polycystic Ovarian Syndrome.
Brief Title: High Intensity Resistance and Aerobic Training Among Women With PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Mobeena Maqsood
Record Dates: First submitted 2022-10-28; First posted 2022-11-02 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Intervention Model Description: Parallel assignment into two groups
Who Masked: Outcomes Assessor
Masking Description: Assessor of this study will be kept blind of the participants treatment group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Resistance Training (Active Comparator): This group will perform high intensity resistance training under supervised physiotherapist in a gym setting. The training load for the first 2 weeks will be 60%-75% of 1RM and increased to 75%-90% of 1RM the following weeks. Load would be increased if the participants will be able to perform 3 sets of 12 repetitions with that load.
  Interventions: Other: High intensity resistance Exercise Training
- High Intensity Aerobic Training (Active Comparator): This group will perform aerobic training under supervision of a physical therapist in gym setting. To calculate exercise intensity, the HR will be maintained at 75-90% of the maximum (HRmax). The training protocol will begin with a 5-minute warm-up and will end with a 5-minute cool down, during which the HR will be 60-75% of the HRmax. At least 90 min of exercise per week for obese PCOS patients, with treadmill walking that may include whole-body movement involving more than 2/3 of the muscles, the exercise intensity will be high intensity
  Interventions: Other: High intensity aerobic Exercise Training

INTERVENTIONS:
Other: High intensity resistance Exercise Training — The resistance training will consist of five resistance exercises (thrice a week on non-consecutive days): squat, leg press, knee extension, lunges, and abdominal crunches. Every participant will be assessed pre and post intervention for hormonal change, BMI/anthropometric measures, fasting glucose and quality of life.The plan will be followed for 12 weeks
  Arms: High Intensity Resistance Training
Other: High intensity aerobic Exercise Training — The training protocol will begin with a 5-minute warm-up and will end with a 5-minute cool down, during which the HR will be 60-75% of the HRmax. At least 90 min of exercise per week for obese PCOS patients, with treadmill walking that may include whole-body movement involving more than 2/3 of the muscles, the exercise intensity will be high intensity
  Arms: High Intensity Aerobic Training

SUMMARY:
polycystic ovarian syndrome (PCOS) is the most common endocrine female disorder, affecting 4-18% women of reproductive age. The prevalence of PCOS in South Asian women, especially in Pakistani women, is much higher (52%) as compared to white population (20 - 25% in UK). On the basis of cultural, environment, diet and lifestyle practices these women are more prone to development of such disorder. So such public health issue needs to be addressed by strong evidence conducted by a clinical trial. The current study is planned to compare effects of two different exercise protocols of high intensity on anthropometric measures, hormonal profile and quality of life.

DETAILED DESCRIPTION:
PCOS is a prevalent condition that is affecting adolescent girls now and has serious impacts on menstrual health and quality of life making them prone to early risk development for chronic metabolic diseases. The comparison between high intensity resistance and aerobic training would give results that which one is more effective in gaining benefits and better effects on overall health both physically(menstrual) as well as mentally that would eventually tell us about the quality of life of such patients.

After the initial screening process, the participants fulfilling the Roterdam criteria, willing to participate in the exercise trial will be recruited and then randomized to the allocated groups of either high intensity resistance or high intensity aerobics. At baseline, their anthropometrics measurements, LH/FSH ratios and fasting plasma glucose test will be done. Patient will be called thrice a week for 3 months for training. It is hypothesized that high intensity resistance or high intensity aerobics will improve anthropometric measures along with hormonal profile and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with PCOS according to Rotterdam criteria
* Age limit: 18-30
* Women who are not part of planned physical activity for the last six months.
* BMI<=30

Exclusion Criteria:

* Women with PCOS who are already on birth control or hormone therapy.
* Women with PCOS who are already are taking some medication for psychological issues
* Women who are already taking cholesterol control medications.
* Women who are a part of any physical activity already

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | changes from Baseline to 4 weeks
  Body mass index (BMI) is a measure of body fat based on height and weight that applies to adult men and women.
Body Mass Index | changes from 4 weeks to 8weeks
  Body mass index (BMI) is a measure of body fat based on height and weight that applies to adult men and women.
Body Mass Index | changes from 8 weeks to 12 weeks
  Body mass index (BMI) is a measure of body fat based on height and weight that applies to adult men and women.
Waist Hip Ratio | changes from Baseline to 4 weeks
  The waist-hip ratio or waist-to-hip ratio (WHR) is the dimensionless ratio of the circumference of the waist to that of the hips
Waist Hip Ratio | changes from 4 weeks to 8weeks
  The waist-hip ratio or waist-to-hip ratio (WHR) is the dimensionless ratio of the circumference of the waist to that of the hips
Waist Hip Ratio | changes from 8 weeks to 12 weeks
  The waist-hip ratio or waist-to-hip ratio (WHR) is the dimensionless ratio of the circumference of the waist to that of the hips
Polycystic ovarian syndrome questionnaire (PCOSQ) | changes from Baseline to 6 weeks
  The PCOSQ consists of five domains, each relating to a common symptom of PCOS; body hair, emotions, infertility, menstrual problems and infertility. Each question on the PCOSQ is associated with a 7-point scale in which 7 represents optimal function and 1 the poorest function.
Polycystic ovarian syndrome questionnaire (PCOSQ) | changes from 6 weeks to 12 weeks
  The PCOSQ consists of five domains, each relating to a common symptom of PCOS; body hair, emotions, infertility, menstrual problems and infertility. Each question on the PCOSQ is associated with a 7-point scale in which 7 represents optimal function and 1 the poorest function.
SF-36 QOL | changes from Baseline to 6 weeks
  The SF-36 is a generic patient-reported outcome measure that quantifies health status and measures health-related quality of life.The SF-36 measures eight scales: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH)
SF-36 Quality of life | changes from 6 weeks to 12 weeks
  The SF-36 is a generic patient-reported outcome measure that quantifies health status and measures health-related quality of life.The SF-36 measures eight scales: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH)

SECONDARY OUTCOMES:
LH/FSH ratios | changes from Baseline to 3 Months
  Luteinizing hormone (LH), follicle-stimulating hormone (FSH), and LH/FSH ratio will be measured when considering a PCOS diagnosis. The LH/FSH ratio is a valid and frequently employed method to test the ovulation and menstrual health of such women and have been reported by many studies

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, Principal Investigator — Riphah International University
Locations (1):
- PostGraduate Lab FRAHS, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benham JL, Booth JE, Corenblum B, Doucette S, Friedenreich CM, Rabi DM, Sigal RJ. Exercise training and reproductive outcomes in women with polycystic ovary syndrome: A pilot randomized controlled trial. Clin Endocrinol (Oxf). 2021 Aug;95(2):332-343. doi: 10.1111/cen.14452. Epub 2021 May 3. PMID 33638879
- [Background] Shele G, Genkil J, Speelman D. A Systematic Review of the Effects of Exercise on Hormones in Women with Polycystic Ovary Syndrome. J Funct Morphol Kinesiol. 2020 May 31;5(2):35. doi: 10.3390/jfmk5020035. PMID 33467251
- [Background] Mario FM, Graff SK, Spritzer PM. Habitual physical activity is associated with improved anthropometric and androgenic profile in PCOS: a cross-sectional study. J Endocrinol Invest. 2017 Apr;40(4):377-384. doi: 10.1007/s40618-016-0570-1. Epub 2016 Oct 22. PMID 27771865
- [Background] Wright PJ, Corbett CF, Pinto BM, Dawson RM, Wirth M. Resistance Training as Therapeutic Management in Women with PCOS: What is the Evidence? Int J Exerc Sci. 2021 Aug 1;14(3):840-854. doi: 10.70252/NEEX8658. eCollection 2021. PMID 34567361
- [Background] Kogure GS, Miranda-Furtado CL, Pedroso DCC, Ribeiro VB, Eiras MC, Silva RC, Caetano LC, Ferriani RA, Calado RT, Dos Reis RM. Effects of Progressive Resistance Training on Obesity Indices in Polycystic Ovary Syndrome and the Relationship With Telomere Length. J Phys Act Health. 2019 Aug 1;16(8):601-607. doi: 10.1123/jpah.2018-0256. PMID 31319405
- [Background] Mitrašinović-Brulić M, Buljan M, Suljević D. Association of LH/FSH ratio with menstrual cycle regularity and clinical features of patients with polycystic ovary syndrome. Middle East Fertility Society Journal. 2021;26(1):40.